CLINICAL TRIAL: NCT05690789
Title: Awareness, Care & Treatment In Obesity Management - An Observation in France
Brief Title: Awareness, Care & Treatment In Obesity Management
Acronym: ACTION-France
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-009; U1111-1267-0332 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- People / Person Living with Obesity (PLwO): From online, general population consumer panels
  Interventions: Other: No treatment given
- Health Care Professionals (HCPs): HCPs treating people who have obesity
  Interventions: Other: No treatment given
- Employers: Single-selection response from defined list
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
ACTION France is a cross-sectional, observational, descriptive, and exploratory survey-based study without collection of laboratory data. The study is not related to any specific treatment options or pharmaceutical product. Collection of data will be performed via quantitative online survey by a third-party vendor.

The goal of this study is to provide insights to drive awareness around the needs of People Living with Obesity (PLwO) and Health Care Professionals (HCPs) involved in obesity treatment and management.

ELIGIBILITY:
Inclusion Criteria:

People Living with Obesity

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, aged above or equal to 18 years at the time of signing informed consent Lives in France
3. Current BMI based on self-reported height and weight of at least 30 kg/m^2

Health Care Professionals

1. Informed consent before any study related activities (study-related activities are any procedure related to recording/collection of data according to protocol)
2. Male or female, aged greater than or equal to 18 years at the time of signing informed consent.
3. Physician with a license to practice
4. Specialty is not surgeon (including bariatric or plastic surgeon)
5. Practices in France
6. In clinical practice greater than or equal to 2 years
7. Spends at least 70 percent time in direct patient care
8. Has seen at least 100 patients in past month
9. Has seen at least 10 patients in past month needing weight management defined as: a patient with a BMI greater than or equal to 30 kg/m^2 with or without comorbidities.

Employers

1. Informed consent before any study related activities (study-related activities are any procedure related to recording/collection of data according to protocol)
2. Age 18 years old or older
3. works in France
4. Company offers health insurance benefits
5. Responsible for making or influencing decisions about employee benefits plan or health and wellness programs
6. works in a company that has at least 20 employees
7. not affiliated with pharma, MR or advertising firms

Exclusion Criteria:

People Living with obesity

1. Previous participation in this study. Participation is defined as having given online consent in this study
2. Currently pregnant
3. Participates in intense fitness or body building programs
4. Has had significant, unintentional weight loss (due to major injury, illness, etc) in the past 6 months
5. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Health Care Providers

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Unwillingness, inability, or language barriers precluding adequate understanding or cooperation.

Employers

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Unwillingness, inability, or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The respondent population will include people living with obesity (PLwO) and health care professionals (HCPs) involved in obesity treatmen, management and employers
Sampling Method: Non-Probability Sample
Enrollment: 1688 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Weight loss motivators | Day 1-day of survey
  Multi-select from defined list
Proportion of PLwO / participants who made serious weight loss effort | Day 1-day of survey
  Percentage of participants
Response to weight loss discussions | Day 1-day of survey
  Single select from defined list
Effective weight loss methods | Day 1-day of survey
  Multi-select from defined list
Obesity attitudes | Day 1-day of survey
  5-point Likert scale
  1=strongly disagree to 5=strongly agree
Attitudes toward prescription weight loss medication and surgery | Day 1-day of survey
  5-point Likert scale
  1=strongly disagree to 5=strongly agree
Weight loss barriers | Day 1-day of survey
  Multi-select from defined list
Obesity and weight management | Day 1-day of survey
  5-point Likert scale
  1=strongly disagree to 5=strongly agree
Degree to which healthcare and society is meeting needs of people living with obesity | Day 1-day of survey
  5-point Likert scale
  1=strongly disagree to 5=strongly agree

SECONDARY OUTCOMES:
Top factors for improving weight loss outcomes | Day 1-day of survey
  Multi-select from defined list
Types of weight management goals | Day 1-day of survey
  Multi-select from defined list
Most helpful information for participants for weight loss | Day 1-day of survey
  Multi-select from defined list
Responsibility for improving health of people living with obesity | Day 1-day of survey
  Multi-select from defined list
Most helpful support for weight loss | Day 1-day of survey
  Multi-select from defined list
Effectiveness of guidelines for treating obesity | Day 1-day of survey
  5-point Likert scale
  1=strongly disagree to 5=strongly agree
Ways participants receive information on weight loss management | Day 1-day of survey
  Multi-select from defined list

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Puteaux, France

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com